CLINICAL TRIAL: NCT05236413
Title: The Effect of a High Fiber Diet and High-Intensity Interval Exercise in Patients With Heart Failure With Preserved Ejection Fraction
Brief Title: The Effect of a High Fiber Diet and High-Intensity Interval Exercise in Patients With HFpEF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: Grain Foods Foundation (Unknown)
Responsible Party: Principal Investigator, Siddartha Angadi, Assistant Professor, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: HSR210393
Record Dates: First submitted 2022-01-31; First posted 2022-02-11 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Heart Failure With Preserved Ejection Fraction
Keywords: HIIT; DASH; High Fiber; HFpEF; heart failure
MeSH Terms: conditions — Heart Failure | interventions — High-Intensity Interval Training; Dietary Approaches To Stop Hypertension; Diet; Exercise

STUDY DESIGN:
Intervention Model Description: Randomized, blinded, 3-arm parallel-group design
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessor will be blinded to group allocations. Subjects will know which group they have been randomized to.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High Intensity Interval Exercise (Experimental): Enrolled patients will perform supervised exercise on 3 nonconsecutive days of the week for 4 weeks.
  Interventions: Behavioral: High Intensity Interval Exercise
- Dietary Approaches to Stop Hypertension (DASH) Diet (Experimental): Enrolled patients will have all of their food prepared for them by a registered dietician for the duration of the study period. The diet will consist of a high fiber content DASH diet.
  Interventions: Behavioral: Dietary Approaches to Stop Hypertension (DASH) Diet
- Exercise + DASH Diet (Experimental): Enrolled subjects will undergo both the exercise training visits and be provided with the DASH diet.
  Interventions: Behavioral: Exercise + DASH Diet

INTERVENTIONS:
Behavioral: High Intensity Interval Exercise — Patients will be required to report for three sessions of supervised stationary cycling exercise per week over a period of 4-weeks. Training heart rates will be determined based on the pre-testing VO2peak and peak heart rate (PHR). All sessions will be supervised by trained personnel.
  Patients will start with eight intervals of 2-min duration at 80-85% of PHR, separated by 2 min of recovery at 50% of PHR, progressing to four, 4-min intervals at 90-95% PHR, separated by 3 min at 50% PHR by the end of week 2.
  Each training session will begin with a 10-min warm-up at 50% of PHR and end with a 5-min cool down at 50% PHR. Subjects will be weighed prior to every exercise session and weight tracked to ensure that their volume status hasn't changed significantly. Subjects will be instructed to maintain usual levels of physical activity and usual diet during the study and not to make any modifications to the same.
  Arms: High Intensity Interval Exercise
Behavioral: Dietary Approaches to Stop Hypertension (DASH) Diet — Patients will be interviewed with regard to their food/religious preferences and food allergies and a 7-day rotating meal plan will be designed per their preferences along with a registered dietitian. This will ensure that patients receive food that is acceptable to them. Participants will then be provided pre-packaged meals for 4-weeks with macronutrient compositions as follows - (Carbohydrates -55-60%, Protein -15-20%, Fat -15-25%, Fiber -35-45g/day). All foods will be labeled, sealed, and packed for weekly delivery and will be designed such that they can be refrigerated or frozen and stored without significant alterations to nutritional content. All food will be prepared by the UVA Hospital Nutrition Services department in conjunction with a registered dietician. Deviations (if any) from the study meal plan will be recorded by the participants in a food record provided at the start of each diet intervention period.
  Arms: Dietary Approaches to Stop Hypertension (DASH) Diet
Behavioral: Exercise + DASH Diet — Patients will undergo both the exercise training intervention and DASH diet as explained above.
  Arms: Exercise + DASH Diet

SUMMARY:
This study is trying to find out how best to improve common measures of health and survival in those diagnosed with heart failure with preserved ejection fraction (HFpEF) through the implementation of 4 weeks of an exercise training program consisting of high intensity interval training, dietary approaches to stop hypertension (DASH diet), or a combination of the two. Currently there are not established guidelines that have been shown to improve clinical end points in those with this HFpEF.

DETAILED DESCRIPTION:
In the face of a rapidly growing population of older, HFpEF patients, there remains a need to identify ideal rehabilitative therapies to enhance improvements in the physical function of these patients. Pharmacological trials in this population have been characterized by a failure to significantly improve exercise tolerance and hard clinical outcomes and this is likely due to their singular cardiovascular focus. Exercise appears to be a promising intervention to improve cardiorespiratory fitness and reduce cardiovascular risk. Further, evidence-based dietary guidelines for patients with heart failure are lacking. Although a high-protein, low-carbohydrate diet is associated with improvements in traditional CV risk markers in patients with heart failure, it may raise cardiovascular risk in this population by adversely affecting endothelial function, increasing susceptibility to myocardial ischemia, and by inducing a pro-inflammatory state due to increased bacterial and LPS translocation through the ischemic gut. Thus, the investigators will explore the effects of the high-carbohydrate, high-fiber DASH diet due to its potential to have salutary effects on vascular risk in this population. In this study, the investigators will examine the singular and combined effects of exercise and a DASH diet in patients with HFpEF on markers of cardiovascular risk.

ELIGIBILITY:
Inclusion Criteria:

* ≥40 years of age
* Diagnosed with heart failure with preserved ejection fraction
* NYHA class II-III symptoms
* Physician clearance to undergo exercise training
* Physician clearance to consume DASH diet
* Complete COVID-19 vaccination status

Exclusion Criteria:

* Unstable angina
* Myocardial infarction in the past 4 weeks
* Uncompensated heart failure
* NYHA class IV symptoms
* Complex ventricular arrhythmias
* Musculoskeletal contraindications to stationary bicycling exercise
* Symptomatic severe aortic stenosis
* Acute pulmonary embolus
* Acute myocarditis
* Uncontrolled hypertension
* Medication non-compliance
* Unable to follow DASH diet
* Food allergies (Nuts, wheat)
* Pregnant women

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
VO2peak | 4 weeks
  Change in VO2peak (L/min) measured pre- and post-intervention

SECONDARY OUTCOMES:
Diastolic Function | 4 weeks
  E' and A' (cm/s) will be used to calculate the E'/A' ratio to assess for diastolic dysfunction and be measured by echocardiogram pre- and post-intervention
Ejection Fraction | 4 weeks
  Ejection fraction (%) will be used to assess changes in cardiac contractile function and be measured by echocardiogram pre- and post-intervention
Global Longitudinal Strain | 4 weeks
  Global longitudinal strain (%) will be used to assess changes in cardiac contractile function and be measured by echocardiogram pre- and post-intervention
Blood pressure | 4 weeks
  Changes in measures of central and brachial blood pressure (mmHg) at pre- and post-intervention
Carotid-Femoral Pulse Wave Velocity | 4 weeks
  Changes in arterial stiffness as measured by carotid-femoral pulse wave velocity (m/s) at pre- and post-intervention
Body Composition | 4 weeks
  Changes in lean and fat mass (grams) will be measured via dual-energy x-ray absorptiometry pre-and post-intervention
Physical Activity Enjoyment Scale | Immediately after the intervention
  Subject enjoyment of exercise will be measured using the Physical Activity Enjoyment Scale. This is an 18 item questionnaire which assess how subjects feel about the exercise they have been performing. Questions are scored using a 7-point likert scale
Minnesota Living with Heart Failure Questionnaire | 4 weeks
  Disease specific quality of life will be measured using the Minnesota Living with Heart Failure Questionnaire (MLHFQ). he MLHFQ consists of 21 items that assess physical and emotional domains. Each item/question is scored on a 0-5 Likert scale.
Epworth Sleepiness Questionnaire | 4 weeks
  The Epworth sleepiness questionnaire is an 8 item questionnaire that measures how likely someone would be to fall asleep in 8 different scenarios. Each item is graded on a 4 point likert scale ranging from "would never nod off" to "high chance of nodding off".
Pittsburgh Sleep Quality Index | 4 weeks
  Sleep quality and sleep disturbances over the pervious month will be measured with the Pittsburgh sleep quality index (PSQI). The PSQI include 19 item self directed questions which look at a measures of sleep quality and a disturbances. It also includes 5 questions to be answered by a roommate (if available) regarding the patients sleep habits.
Circadian Type Questionnaire | 4 weeks
  The Circadian Type Questionnaire is an 19 item VAS that is used to assess someones ability to change their sleeping habits.
Sleep Apnea | 4 weeks
  Changes in sleep apnea will be measured using a WatchPAT device. This device measured finger peripheral arterial tone and measures arterial volume changes in the finger. This reflect changes in sympathetic tone and is associated with sleep disordered breathing.

OTHER OUTCOMES:
NTproBNP | 4 weeks
  Assess changes in NTproBNP (pg/ml) as a biomarker of myocardial strain at pre- and post-intervention
Inflammation | 4 weeks
  C-reactive protein (mg/dl) will be used as a biomarker for inflammation to be measured pre- and post-intervention
Lipids | 4 weeks
  A lipid panel will be performed to measure total cholesterol, triglycerides, high-density lipoproteins, and low-density lipoprotein (mg/dl) to assess changes in cardiometabolic health pre- and post-intervention
Insulin | 4 weeks
  Fasting insulin levels (U/ml) will be tested to assess changes in cardiometabolic health pre- and post-intervention
Fasting Blood Glucose | 4 weeks
  Fasting blood glucose levels (mg/dl) will be tested to assess changes in cardiometabolic health pre- and post-intervention
Endothelin-1 | 4 weeks
  Arterial vasoconstrictor tone will be assessed by serum endothelin-1 (pg/mL) at pre- and post-intervention.
Lipopolysaccharide | 4 weeks
  Gut mucosal health and inflammation as measured by plasma Lipopolysaccharides (ng/mL) pre- and post-intervention
Trimethylamine-N-oxide | 4 weeks
  Trimethylamine-N-oxide (µM) will be used to assess gut mucosal health and inflammation pre- and post-intervention

CONTACTS AND LOCATIONS:
Overall Officials: Siddhartha S Angadi, PhD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia University Hospital, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No
Deidentified data will be shared on request.